CLINICAL TRIAL: NCT01310881
Title: A Phase 1, Randomized, Subject Single Blinded, Placebo-Controlled, Single-Dose Escalation Study Evaluating the Safety, Tolerability, and Pharmacokinetics (PK) of NSI-189 Phosphate in Healthy Subjects
Brief Title: Single-Dose Pharmacokinetics (PK) Study of Novel Neurogenic Compound NSI-189
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS2010-2
Record Dates: First submitted 2011-02-24; First posted 2011-03-09 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-05

CONDITIONS: Depression
Keywords: Neurogenesis; hippocampal stem cells; depression; stroke
MeSH Terms: conditions — Depression; Stroke | interventions — NSI-189

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Dose 1 (Experimental)
  Interventions: Drug: NSI-189 Phosphate
- Dose 2 (Experimental)
  Interventions: Drug: NSI-189 Phosphate
- Dose 3 (Experimental)
  Interventions: Drug: NSI-189 Phosphate
- Dose 4 (Experimental)
  Interventions: Drug: NSI-189 Phosphate
- Dose 5 (Experimental)
  Interventions: Drug: NSI-189 Phosphate
- Dose 6 (Experimental)
  Interventions: Drug: NSI-189 Phosphate
- Dose 7 (Experimental)
  Interventions: Drug: NSI-189 Phosphate

INTERVENTIONS:
Drug: NSI-189 Phosphate — Once daily oral administration

SUMMARY:
This is a subject single blinded, randomized, placebo-controlled, single dose, first-time-in-human study with three or more ascending cohorts.

DETAILED DESCRIPTION:
Each subject will undergo Screening (Day -28 to Day -2). Subjects will return to the clinical site on Day -1, be admitted to the unit, and eligibility will be reconfirmed. Eligible subjects will receive a single dose of investigational medicinal product (IMP, NSI-189 Phosphate or Placebo) on Day 1 and will be followed for safety and PK until discharge on Day 3. Subjects who are experiencing any significant AEs that are considered possibly related to study drug will be kept at the unit for an additional day (or longer) until the event resolves or it is considered medically safe for the subject to be discharged. Subjects will have a telephone Follow-up on Day 4 and return to the unit on Day 7 (± 1) for End-of-study. Participation of an individual subject may last up to 36 days from the time of Screening until the End-of-study.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet all of the following criteria:

  1. Subject has the ability to understand the purpose and risks of the study and to provide signed and dated informed consent.
  2. Males and females between 18 to 55 years of age, inclusive, at the time of informed consent.
  3. The following applies to female subjects:

     • Non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year with follicle stimulating hormone >40 U/L).
  4. The following applies to male subjects:

     • Male subjects with a female partner of childbearing potential will be required to use an effective method of birth control or practice abstinence during this study and for 3 months following discontinuation of IMP.
  5. Non-smokers (or other nicotine use) as determined by history (no nicotine use over the past year) and by negative urine cotinine test at screening and Day -1.
  6. BMI ≥ 19.5 and ≤30.0 kg/m2, at screening. Bodyweight must be >50 kg.
  7. Healthy, determined by pre-study medical evaluation and investigator discretion (medical history, physical examination, vital signs, ECG, and clinical laboratory evaluations).

Exclusion Criteria:

1. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, dermatological or psychiatric disorder(s), or other major disease as determined by the Investigator or designee.
2. History of seizures including febrile seizures, loss of consciousness, or any clinically significant finding on the neurologic examination.
3. Clinically significant abnormal clinical chemistry values, as determined by the Investigator.
4. Clinically significant (as determined by the Investigator) 12-lead ECG abnormalities, including corrected QT interval using Bazett's correction method of >450 msec for males and >470 msec for females.
5. History of severe allergic or anaphylactic reactions.
6. Subjects who have plans to undergo elective procedures/surgeries at any time during the study through the follow-up visits.
7. A positive screening test for human immunodeficiency virus (HIV), hepatitis C virus antibody (HCVAb), hepatitis B core antibody (HBcAb), or hepatitis B surface antigen (HBsAg).
8. Serious infection (e.g. pneumonia, septicemia) as determined by the Investigator within 3 months prior to Day -1.
9. Fever or bacterial, or viral infection (including upper respiratory tract infection) within 2 weeks prior to Day -1.
10. Treatment with any prescribed medication within 28 days prior to Day -1.
11. Treatment with any over-the-counter products (OTC), including herbal and/or alternative health preparations and procedures within the 14 days prior to Day -1. Note: Intermittent treatment with acetaminophen [≤1000 mg/day] and/or ibuprofen [≤400 mg/day] is permitted.
12. Current enrollment in any other drug, biologic, device, or clinical study, or treatment with an investigational product or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) prior to Day -1.
13. Any live or attenuated immunization/vaccination within 1 month prior to the study drug administration or planned to occur during the study period.
14. Donation of blood (>500 mL) or blood products within 1 month prior to screening.
15. History of alcohol or substance abuse (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, etc.) (as determined by the Investigator).
16. Vigorous exercise (as determined by the Investigator) within 48 hours prior to the study drug administration.
17. Inability to comply with study requirements.
18. Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
19. Any concurrent disease or condition that, in the opinion of the Investigator, would make the subject unsuitable for participation in the clinical study.
20. Subject unwilling to avoid consumption of coffee and caffeine containing beverages within 48 hours prior to Day -1 until discharge from the clinical site.
21. Use of an investigational product within 30 days prior to Day -1.
22. Subject is unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study.
23. Subject is unlikely to comply with the protocol requirements, instructions and study-related restrictions.
24. Subject has previously been enrolled in this clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety of drug assessed by number and severity of adverse events in drug vs placebo groups | 7 days
  Values for vital signs, standard physical examination, ECG, EEG and standard clinical laboratory tests (haematology and biochemistry), and for standard neurological exam and the Columbia Suicide Severity Rating Scale will be compared between NS189 and placebo.

SECONDARY OUTCOMES:
Pharmacokinetics of NS189 will be determined by plasma sample collection at various timepoints post-dosing, and measuring concentration of drug over time. | 7 days
  Concentration of NS189 will be measured in plasma and standard PK values determined: AUC, Cmax, Tmax, T1/2, CL, Vz

CONTACTS AND LOCATIONS:
Overall Officials: Karl Johe, PhD, Study Director — Neuralstem Inc.; David Han, MD, Principal Investigator — California Clinical Trials
Locations (1):
- California Clinical Trials, Glendale, California, United States

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Deng W, Aimone JB, Gage FH. New neurons and new memories: how does adult hippocampal neurogenesis affect learning and memory? Nat Rev Neurosci. 2010 May;11(5):339-50. doi: 10.1038/nrn2822. Epub 2010 Mar 31. PMID 20354534
- [Background] DeCarolis NA, Eisch AJ. Hippocampal neurogenesis as a target for the treatment of mental illness: a critical evaluation. Neuropharmacology. 2010 May;58(6):884-93. doi: 10.1016/j.neuropharm.2009.12.013. Epub 2010 Jan 6. PMID 20060007
- [Background] Marlatt MW, Lucassen PJ. Neurogenesis and Alzheimer's disease: Biology and pathophysiology in mice and men. Curr Alzheimer Res. 2010 Mar;7(2):113-25. doi: 10.2174/156720510790691362. PMID 19860727
- [Background] Kernie SG, Parent JM. Forebrain neurogenesis after focal Ischemic and traumatic brain injury. Neurobiol Dis. 2010 Feb;37(2):267-74. doi: 10.1016/j.nbd.2009.11.002. Epub 2009 Nov 10. PMID 19909815
- [Background] Kempermann G, Krebs J, Fabel K. The contribution of failing adult hippocampal neurogenesis to psychiatric disorders. Curr Opin Psychiatry. 2008 May;21(3):290-5. doi: 10.1097/YCO.0b013e3282fad375. PMID 18382230